CLINICAL TRIAL: NCT06288763
Title: Nerve Transfer to Restore Upper Limb Function and Quality of Life in High Tetraplegia
Brief Title: Nerve Transfer to Improve Function in High Level Tetraplegia
Status: Recruiting | Type: Observational
Sponsor: Wilson Z. Ray (Other)
Collaborators: University of Michigan (Other); The Methodist Hospital Research Institute (Other); University of Pennsylvania (Other); University of Utah (Other); Stanford University (Other); University of Miami (Other); Johns Hopkins University (Other); University of Alberta (Other); Wake Forest University Health Sciences (Other); Department of Defense / Congressionally Mandated Research Program (CDMRP) (Unknown)
Responsible Party: Sponsor-Investigator, Wilson Z. Ray, MD - Principal Investigator, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: CDMRP-eBRAP-SC220192
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cervical Spinal Cord Injury; Tetraplegia
Keywords: Spinal Cord Injury; Cervical spinal cord injury; Nerve Transfer Surgery; High Cervical Spinal Cord Injury; Cervical SCI; Tetraplegia; Quadriplegia; Nerve transfer; Spinal Accessory Nerve
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine if nerve transfer surgeries improve upper extremity function and quality of life in patients with a high level cervical spinal cord injury.

Participants will:

* undergo standard of care pre- and post-op testing and study exams
* complete pre- and post-questionnaires
* undergo standard of care nerve transfer surgeries
* follow-up with surgeon at 6/12/18/24/36 and potentially at 48 months
* attend therapy at local therapist for up to 2 years postop.

DETAILED DESCRIPTION:
Restoration of function in patients with high tetraplegia has been an elusive clinical challenge. There is a critical need to find an effective reconstructive therapy/procedure which improves the upper extremity function in patients with high tetraplegia.

One pure motor nerve - spinal accessory nerve (SAN) remains a viable donor in high tetraplegia patients to successfully restore elbow flexion or extension. Elbow function can provide profound independence in mobility, ventilator management and may broaden the application of assistive therapies.

The two objectives of this study are:

* Determine if SAN nerve transfer surgery can improve the reinnervation of bicep or tricep muscles in high tetraplegia patients.
* Determine if SAN nerve transfer surgery can reanimate upper arm function and improve functional independence in patients with high tetraplegia.

Study Activities (including standard of care (SOC))

* Electrodiagnosis pre-op (SOC)
* Upper extremity maximum muscle testing (SOC)
* Questionnaires (SOC and study-related (SR))
* Exams by a study therapist (SR)
* Neurological exam - ISNCSCI - (SOC)
* Nerve Transfer Surgery to be determined by surgeon (SOC)
* Follow-up visits with surgeon at 6/12/18/24/36 and potentially 48 months
* post-op electrodiagnostic testing (SR)
* post-op upper extremity maximum muscle testing (SOC)
* post-op questionnaires
* post-op therapy exams (SR)

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* High cervical SCI (motor level C1-C4)
* Motor complete SCI AIS grade A-B
* Plateaued spontaneous recovery for at least 6 months of non-operative therapy
* SCI greater than 6 months and fewer than 60 months since injury
* At least MRC 4/5 donor strength
* Mentally and physically willing and able to comply with evaluations

Exclusion Criteria:

* Active infection at the operative site or systemic infection
* Any return or ongoing recovery of distal motor function
* Significant joint contractures and/or limitations in passive range of motion in the arm
* Mentally or physically compromised making it impossible to complete study activities
* Immunologically suppressed
* Currently undergoing long-term steroid therapy
* Active malignancy
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-level SCI injury (C1-C4) with complete lack of upper extremity function. Occurrence of injury should be greater than 6 months but fewer than 60 months
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Elbow Dynamometry | 36-48 months post-surgery
  Change from baseline to 36-48 months post-surgery. Elbow dynamometer measures muscle strength using a handheld portable dynamometer
Spinal Cord Independence Measure | 36-48 months post-surgery
  Change from baseline to 36-48 months post-surgery. SCIM addresses three specific areas of function in patients with SCI, 1) Self-care (feeding, grooming, bathing, and dressing), 2) respiration and sphincter management, and 3) patient's mobility abilities (transfers from bed and indoors/outdoors). SCIM guide clinicians in determining treatment goals/objectives for SCI patients helping therapists assess measurable outcomes in their functional independence. Scores range from 0-100 with a higher score representing better function.
Motor strength in medical research council grade (MRC) | 36-48 months post-surgery
  Change in baseline to 36-48 Months post-surgery. The manual muscle testing is a reliable measure of motor strength when assessed by a trained examiner. Scores range from 0-5, with the highest number representing a better score.
Electrodiagnosis (Nerve Conduction Study and Electromyography | 36-48 months post-surgery
  Change in baseline to 36-48 Months post-surgery. NCS/EMG evaluate neuromuscular health and inform the integrity of lower motor neurons.

SECONDARY OUTCOMES:
Canadian Outcomes Performance Measure (COPM) | 36-48 Months post-surgery
  Change from baseline to 36-48 months post-surgery. COPM is a validated outcome measure for SCI patients focusing on occupational performance in all areas of life. Scores range from 5-50 for performance and satisfaction. The higher scores reflect better performance and satisfaction.
Capabilities of Upper Extremity Questionnaire (CUE-Q) | 36-48 Months post-surgery
  Change from baseline to 36-48 months post-surgery. CUE-Q detects changes in upper extremity function. Scores range from 32-224 with higher scores reflecting better function.
Modified Ashworth Scale (MAS) | 36-48 Months post-surgery
  Change from baseline to 36-48 months post-surgery. MAS is a reliable measure for rating spasticity in SCI. Scores range from 0-32 with higher scores reflecting better function.
Spinal Cord Injury Quality of LIfe Questionnaire | 36-48 Months post-surgery
  Change from baseline to 36-48 months post-surgery. SCI-QOL is designed to measure subjective quality of life in terms of satisfaction and importance. Range of scores is 0 to 30 with the higher scores reflecting a better quality of life..
International SCI Pain Basic Dataset (ISCIPBDS) | 36-48 Months post-surgery
  Change from baseline to 36-48 months post-surgery. ISCIPBDS correctly classifies pain, determines its intensity and broad impact on daily activities. Lower scores reflect less pain/less interference in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Z. Ray, MD, Principal Investigator — Washington University School of Medicine
Locations (10):
- United States (9):
  - Stanford University, Stanford, California
  - University of Miami, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared

REFERENCES:
- See also: Washington University Neurosurgery Website — http://www.neurosurgery.wustl.edu